CLINICAL TRIAL: NCT00626522
Title: A Randomised, 4-week, Placebo-controlled, Double-blind, 6 Arm Parallel Group, Dose-finding Clinical Trial, to Assess the Efficacy, Safety and Pharmacokinetics of Three Different Doses of Formoterol Combined With the Inhaled Anticholinergic Aclidinium Bromide, Aclidinium Bromide Monotherapy and Formoterol Monotherapy All Administrated Once Daily by Inhalation Via Almirall Inhaler in Patients With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease.
Brief Title: Aclidinium/Formoterol Fixed Combination Dose Finding Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M/273FO/23; 2007-004435-30 (EudraCT Number)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Bronchitis; Chronic; Emphysema; Smokers or ex-Smokers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Bronchiolitis Obliterans Syndrome; Emphysema; Smoking Cessation | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: Aclidinium bromide and formoterol
- 2 (Experimental)
  Interventions: Drug: Aclidinium bromide and formoterol
- 3 (Experimental)
  Interventions: Drug: Aclidinium bromide and formoterol
- 4 (Placebo Comparator)
  Interventions: Drug: Aclidinium bromide and formoterol placebo
- 5 (Placebo Comparator)
  Interventions: Drug: Aclidinium bromide and formoterol placebo
- 6 (Placebo Comparator)
  Interventions: Drug: Aclidinium bromide and formoterol placebo

INTERVENTIONS:
Drug: Aclidinium bromide and formoterol — once daily
  Arms: 1; 2; 3
Drug: Aclidinium bromide and formoterol placebo — once daily
  Arms: 4; 5; 6

SUMMARY:
The study seeks to determine the optimal dose of the Aclidinium/Formoterol combination for investigation in Phase III clinical trials

DETAILED DESCRIPTION:
Dose-finding clinical trial, to assess the efficacy, safety and pharmacokinetics of three different doses of formoterol combined with the inhaled anticholinergic aclidinium bromide, aclidinium bromide monotherapy and formoterol monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or non-pregnant, non-lactating females aged between 40 and 80 years old, both inclusive. Women of childbearing potential were allowed to enter the trial only if they used two medically approved contraceptive measures (ie, mechanical and pharmacological).

   (A female was considered to be of childbearing potential unless she had a hysterectomy, was at least one year post-menopause or had undergone tubal ligation. All women of childbearing potential were to have a negative serum pregnancy test at the Screening Visit).
2. Patients with a clinical diagnosis of stable moderate to severe COPD (stages II and III) according to the GOLD 2006 classification (http://www.goldcopd.com).
3. Current or ex-cigarette smoker with a smoking history of at least 10 pack-years.

   Pack-years were calculated by dividing the number of cigarettes smoked per day by 20 (the number of cigarettes in a pack) and multiplying this figure by the number of years a person had smoked. For example, a person who smoked 40 cigarettes a day and had smoked for 10 years would have had a 20 pack-year smoking history (40 cigarettes per day ÷ 20 cigarettes per pack = 2; 2 x 10 years of smoking = 20 pack-year history).

   Patients smoking other tobacco types were not allowed, unless they met the cigarette criterion as well.
4. Patients whose Forced Expiratory Volume in 1 second (FEV1) at the Screening Visit measured between 30-45 minutes post inhalation of 400 μg of salbutamol was 30% ≤FEV1 <80% of the predicted normal value (ie, 100 x Post-salbutamol FEV1/Predicted FEV1 <80% and ≥30%). (Predicted normal values used for calculation purposes were to be based on European Community for Steel and Coal predicted values)
5. Patients whose FEV1/Forced Vital Capacity (FVC) at the Screening Visit measured between 30- 45 minutes post inhalation of 400 μg of salbutamol was <70% (ie, 100 x Post-salbutamol FEV1/FVC <70%).
6. Patients whose COPD symptoms and FEV1 values at the time of randomisation were stable compared to the Screening Visit, according to the Investigator's medical judgment.
7. Patients who were eligible and able to participate in the trial and who consented to do so in writing after the purpose and nature of the investigation had been explained.

Exclusion Criteria:

1. History or current diagnosis of asthma, allergic rhinitis or atopy, or exercise-induced bronchospasm.
2. Eosinophil count ≥600 cells/mm3.
3. Clinically significant respiratory conditions at the time of Screening Visit defined as:

   * Use of long-term oxygen therapy >5 h/day,
   * Known active tuberculosis,
   * History of interstitial lung or pulmonary thromboembolic disease,
   * Pulmonary resection during the past 12 months,
   * History of life-threatening COPD,
   * History of bronchiectasis secondary to respiratory diseases others than COPD (eg, cystic fibrosis, Kartagener's syndrome, etc),
   * Patients who in the Investigator's opinion may have needed to stop or start pulmonary rehabilitation or undergo a thoracotomy during the trial,
4. Hospitalisation due to COPD exacerbation, up to the 3 months prior to the Screening Visit.
5. Signs of a COPD exacerbation or respiratory infection (including the upper respiratory tract), up to the 6 weeks prior to the Screening Visit.
6. Clinically significant cardiovascular conditions at the time of Screening Visit defined as:

   * Myocardial infarction within the previous 6 months,
   * Unstable arrhythmia which has required changes in the pharmacological therapy or other intervention within the previous 12 months, or newly diagnosed arrhythmia within the previous 3 months.
   * Hospitalisation within the previous 12 months for heart failure functional classes III (marked limitation of activity and only comfortable at rest) and IV (need of complete rest, confinement to bed or chair, discomfort at any physical activity and presence of symptoms at rest) as per the New York Heart Association classification (www.americanheart.org)
   * Thoracic surgery within the previous 24 months
7. Presence of symptomatic prostatic hypertrophy and/or bladder neck obstruction. (However, patients who had a diagnosis of these conditions but without symptoms due to stable concomitant medication for its treatment were allowed to enter trial).
8. Presence of narrow-angle glaucoma.
9. History of untoward reactions or known hypersensitivity to inhaled anticholinergics (including aclidinium bromide), β2 adrenergic agonists or inhaled medication or any component thereof (including report of paradoxical bronchospasm).
10. Life expectancy of less than 1 year.
11. Prolonged QT interval corrected using Bazett's formula (QTcB) interval (>470 msec) in any of the ECGs performed before randomisation, and/or the use of drugs which may have induced its prolongation.
12. Clinically relevant abnormalities in laboratory results, ECG parameters (other than QTcB), or physical examination if the abnormality defines a disease state listed as an exclusion criterion, except for those related to COPD.
13. Clinically significant diseases other than COPD, which, in the opinion of the Investigator, may have put the patient at risk because of the participation in the trial; or diseases which may have influenced the results of the study or the patient's ability to take part in it.
14. Patients who did not maintain regular day/night, waking/sleeping cycles (eg, night shift workers were to be excluded).
15. Patients who intended to use any concomitant medication not permitted by the protocol or who had not undergone the required wash-out period for a particular prohibited medication.
16. Patients who were unable or unlikely to be cooperative with the study requirements of taking the medication, completion of the Patient Diary and attending the clinic for study visits.
17. Patients who were unable to properly use a dry powder or pressurised metered-dose inhalers (pMDI) inhaler device and/or to perform acceptable and reproducible spirometry measurements as per the ATS/ERS standards (Standardisation of lung function test, 2005 20).
18. History of drug and/or alcohol abuse or addiction during the previous 2 years.
19. Previous participation in another clinical trial with any investigational medicinal product 6 weeks prior to the Screening Visit. (Patients who had participated in a previous clinical trial with aclidinium bromide (Almirall product code LAS34273) were to be allowed to participate in this study provided that the above criterion was fulfilled. This circumstance was to be specifically recorded on the eCRF).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (9):
- Australia (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Research Site, Moscow, Czechia
- Poland (2):
  - Research Site, Saint Petersburg
  - Research Site, St-Petersburg
- Russia (4):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Yaroslavl

REFERENCES:
- See also: Sponsor website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp
- See also: Co-Sponsor website — http://www.frx.com/
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3953&filename=Synopsis-m-273FO-23-Final.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a total of 81 sites: 21 in Russia, 13 in Poland, 8 in India, 8 in Romania, 6 in Australia, 5 in Taiwan, 5 in the Czech Republic, 5 in New Zealand, 4 in Hungary, 3 in Malaysia and 3 in Slovakia
  The first patient was screened in February 2008 and the last patient visit was in November 2008
Pre-assignment Details: A total of 808 patients were screened and 566 were randomized into the study
  Among 242 patients who failed to be randomized, the main reason for screen failure was non-fulfillment of one or more study entry criteria (156 patients), followed by subject's personal request (32 patients)
Groups:
- Aclidinium 200 μg / Formoterol 6 μg: Aclidinium bromide 200 μg + formoterol fumarate 6 μg fixed dose combination (FDC) once-daily
- Aclidinium 200 μg / Formoterol 12 μg: Aclidinium bromide 200 μg + formoterol fumarate 12 μg fixed dose combination (FDC) once-daily
- Aclidinium 200 μg / Formoterol 18 μg: Aclidinium bromide 200 μg + formoterol fumarate 18 μg fixed dose combination (FDC) once-daily
- Aclidinium 200 μg: Aclidinium bromide 200 μg once-daily
- Formoterol 12 μg: Formoterol fumarate 12 μg once-daily
- Placebo: Placebo once-daily
Period: Overall Study
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Started | 121 | 120 | 125 | 76 | 65 | 59
Completed | 115 | 113 | 117 | 74 | 58 | 57
Not Completed | 6 | 7 | 8 | 2 | 7 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 5 | 5 | 0 | 4 | 1
Not completed — COPD exacerbation | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Inconsistent reason reported | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-fulfilment of in/exclusion criteria | 1 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo | Total
Number analyzed (Participants) | 121 | 120 | 125 | 76 | 65 | 59 | 566
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (9.0) | 63.6 (8.9) | 63.9 (8.1) | 63.7 (9.3) | 64.0 (9.8) | 60.7 (7.8) | 63.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 29 | 16 | 11 | 15 | 123
  Male | 91 | 98 | 96 | 60 | 54 | 44 | 443

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) for 0-12 hr
Time Frame: Baseline and treatment Week 4
Population: ITT Population defined as all randomised patients who took at least one dose of investigational medicinal product and had at least the baseline and one post-baseline efficacy assessments
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 112 | 111 | 115 | 71 | 54 | 55
Liters | 0.170 [0.128 to 0.213] | 0.219 [0.176 to 0.262] | 0.230 [0.187 to 0.273] | 0.075 [0.021 to 0.129] | 0.099 [0.037 to 0.161] | -0.036 [-0.097 to 0.025]
Statistical Analysis 1: Comparison: Aclidinium 200 μg / Formoterol 6 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares mean difference = 0.206, 95% CI 2-sided [0.131 to 0.280], Standard Error of Mean 0.038
Statistical Analysis 2: Comparison: Aclidinium 200 μg / Formoterol 12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares mean difference = 0.254, 95% CI 2-sided [0.180 to 0.329], Standard Error of Mean 0.038
Statistical Analysis 3: Comparison: Aclidinium 200 μg / Formoterol 18 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least squares mean difference = 0.265, 95% CI 2-sided [0.191 to 0.340], Standard Error of Mean 0.038

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline and treatment Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 117 | 117 | 121 | 73 | 63 | 56
Liters | 0.042 [0.001 to 0.084] | 0.085 [0.044 to 0.127] | 0.044 [0.003 to 0.085] | -0.017 [-0.70 to 0.036] | 0.014 [-0.043 to 0.071] | -0.031 [-0.091 to 0.029]

3. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline and treatment Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 121 | 120 | 124 | 75 | 65 | 58
Liters | 0.294 [0.250 to 0.338] | 0.357 [0.313 to 0.401] | 0.349 [0.305 to 0.393] | 0.184 [0.128 to 0.240] | 0.216 [0.156 to 0.276] | 0.044 [-0.019 to 0.108]

4. Secondary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) for 0-3 hr
Time Frame: Baseline and treatment Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 121 | 120 | 124 | 75 | 65 | 56
Liters | 0.197 [0.158 to 0.236] | 0.256 [0.217 to 0.295] | 0.250 [0.211 to 0.289] | 0.088 [0.038 to 0.138] | 0.134 [0.081 to 0.188] | -0.033 [-0.091 to 0.024]

5. Secondary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) for 0-6 hr
Time Frame: Baseline and treatment Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 115 | 112 | 115 | 72 | 56 | 55
Liters | 0.206 [0.164 to 0.249] | 0.266 [0.223 to 0.309] | 0.272 [0.229 to 0.314] | 0.094 [0.040 to 0.148] | 0.137 [0.076 to 0.198] | -0.033 [-0.094 to 0.029]

ADVERSE EVENTS:
Time Frame: Up to Day 38
Arm/Group | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 18 μg | Aclidinium 200 μg | Formoterol 12 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/121 | 1/120 | 3/125 | 0/76 | 1/65 | 0/59
Other Adverse Events (participants affected / at risk) | 2/121 | 1/120 | 3/125 | 4/76 | 5/65 | 2/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium 200 μg / Formoterol 6 μg (N=121) | Aclidinium 200 μg / Formoterol 12 μg (N=120) | Aclidinium 200 μg / Formoterol 18 μg (N=125) | Aclidinium 200 μg (N=76) | Formoterol 12 μg (N=65) | Placebo (N=59)
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive pulmonary disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium 200 μg / Formoterol 6 μg (N=121) | Aclidinium 200 μg / Formoterol 12 μg (N=120) | Aclidinium 200 μg / Formoterol 18 μg (N=125) | Aclidinium 200 μg (N=76) | Formoterol 12 μg (N=65) | Placebo (N=59)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 4 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and/or presentation whether complete or partial, of any part of the data or results of this trial, will be subject to revision and written agreement between the investigator and sponsor.